CLINICAL TRIAL: NCT02960126
Title: Comparison of Efficacy and Safety Between Aspirin and Clopidogrel in the Atrial Fibrillation With Low or Moderate Stroke Risk
Brief Title: Efficacy and Safety of Aspirin and Clopidogrel in the Atrial Fibrillation With Low or Moderate Stroke Risk
Acronym: CESAC-AF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Sang Min Park, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CESAC-AF
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Clopidogrel (Active Comparator): Case management with clopidogrel 75mg once daily is provided for stroke prevention in AF patient.
  Interventions: Drug: Clopidogrel
- Control: Aspirin (Experimental): Usual care with aspirin 100mg once daily is provided for stroke prevention in AF patient.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin
  Arms: Control: Aspirin
Drug: Clopidogrel
  Arms: Intervention: Clopidogrel

SUMMARY:
This study was designed in order to evaluate and compare the efficacy and safety between aspirin and clopidogrel in the patient with low stroke risk Atrial Fibrillation (AF).

DETAILED DESCRIPTION:
Efficacy outcome will be evaluated the major cerebro-cardiovascular event including stroke, cardiovascular death, and myocardial infarction during 1 year-medication period. In addition, safety outcome will be evaluated the gastrointestinal responses including peptic ulcer and upper gastrointestinal bleeding events to both study drugs by repeated gastroenteroscopic examinations before and after medication by GI specialist.

ELIGIBILITY:
Inclusion Criteria:

1. Man or Women > 20 years old
2. newly detected AF (CHA2DS2VASc index score: 1)
3. Patient who needs antiplatelet therapy using aspirin clopidogrel for stroke prevention
4. volunteer only
5. childbearing aged women who takes proper oral contraceptive

Exclusion Criteria:

1. No specific contraindication or any history of hypersensitivity of Clopidogrel or aspirin
2. Patient with active GI bleeding or bleeding tendency or major bleeding history
3. less than 1 year of residual expected life
4. Pregnant or breast-feeding women
5. Other causes, determined by charged physician
6. Patient with definite GERD who needs special treatment
7. Patient who needs to take NSAID (Non-Steroidal Anti-Inflammatory Drug) for more than 2 weeks

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Major Cerebrovascular and cardiac events including stroke, CV death, MI | 1 year after randomization
  Number of each event
Major gastrointestinal event including peptic ulcer disease and bleeding | 1 year after randomization
  Number of each event

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SM, Jeong H, Jung MH, Hong KS, Hong MK, Bang CS, Kim CY. Rationale and Design for a Randomized Comparison of Efficacy and Safety between Aspirin and Clopidogrel in Atrial Fibrillation Patients with Low Stroke Risk: CESAC-AF trial. Contemp Clin Trials. 2017 Sep;60:51-55. doi: 10.1016/j.cct.2017.06.011. Epub 2017 Jun 19. PMID 28642210